CLINICAL TRIAL: NCT05664828
Title: A Phase IIa, Single Centre, Open Label, Proof of Concept Study Concerning Efficacy of the Novel Intravenous Contrast Agent SN132D in Patients With Suspected Endometriosis.
Brief Title: Efficacy of SN132D in Patients With Suspected Endometriosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spago Nanomedical AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SPAGOPIX-02; 2022-000652-11 (EudraCT Number)
Record Dates: First submitted 2022-12-07; First posted 2022-12-27 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2022-12

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Intervention Model Description: Open-label, non-randomised and non-placebo-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single dose (i.v.) SN132D (Experimental): SN132D is a nanoparticle solution at 20 µmol Mn/kg dosage, administrated via intravenous infusion.
  Interventions: Drug: SN132D

INTERVENTIONS:
Drug: SN132D — Manganese-based macromolecular MRI contrast agent
  Other Names: SpagoPix

SUMMARY:
This is a Phase IIa, open-label, non-randomised and non-placebo-controlled study. The study is designed to evaluate the diagnostic value and safety of a single intravenous dose of SN132D in up to 18 participants with suspected endometriosis. Magnetic resonance imaging (MRI) will be performed pre- and post-infusion of SN132D.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent including willingness to undertake 3 MRI investigations in one day.
2. Females with endometriosis or suspected endometrial lesions at transvaginal ultrasound examination.
3. At least 18 years of age when signing the informed consent.
4. Adequate renal and hepatic function:

   eGFR ≥ 50 mL/min/1.73 m2, bilirubin <1 x upper limit of normal (ULN), creatinine <1 x ULN, ASAT and ALAT < 1 x ULN, Bilirubin ULN: 25 µmol/L, creatinine ULN: 90 µmol/L, ASAT ULN: 0.60 µkat/L and ALAT ULN: 0.75 µkat/L) at the screening visit.
5. Females of child-bearing potential* must agree to the use of effective contraception** or practice abstinence during the study and for 30 days after the IMP administration.

   *A female of child-bearing potential is a sexually mature female who 1) has not undergone a hysterectomy or bilateral oophorectomy, or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e. had had menses at any time in the preceding 24 consecutive months).

   **Effective contraception is defined as contraceptive methods with a failure rate of < 1% to prevent pregnancy (combined [oestrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD]or intrauterine hormone-releasing system [IUS]).
6. Adequate haematological function: haemoglobin (Hb) ≥90 g/L, absolute neutrophil count (ANC) ≥1.3x109 /L and platelet count ≥ 100 x 109 /L.

Exclusion Criteria:

1. Female participants who are pregnant or who are currently breast feeding.
2. Conditions contraindicating MRI including, but not limited to, BMI > 40 kg/m2 at screening claustrophobia, metallic implants or internal electrical devices (e.g., cochlear implant, nerve stimulator, gastric pacemaker, bladder stimulator, pacemaker, defibrillator, artificial valves in heart, aneurysm clips, etc.), and permanent makeup or tattoos which in the Investigator's opinion might jeopardise the patient's safety or interfere with the imaging measurements. The Investigator is encouraged to contact the MR clinic for advice on which implants, tattoos, etc may be unsuitable.
3. Moderate to severe hypertension as judged by the Investigator.
4. History of significant cardiovascular disease such as myocardial infarction, congestive heart failure, stroke, serious cardiac arrhythmias, history of angina within 6 months prior to screening.
5. Clinically diagnosed obstruction of bile duct as judged by the Investigator.
6. Electrocardiogram (ECG) abnormalities in the standard 12-lead ECG (at screening) which, in the opinion of the Investigator is clinically relevant, or will interfere with the ECG analysis.
7. Abnormalities detected during examination at screening and admission, which in the opinion of the Investigator, may either put the patient at risk because of participation in the study or influence the results or the patient's ability to participate in the study.
8. Active infection requiring systemic treatment within one week prior to agent administration.
9. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the results or the patient's ability to participate in the study.
10. Known human immunodeficiency virus (HIV) infection, active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection requiring treatment. Participants with chronic HBV or HCV infection are eligible at the Investigator's discretion provided that the disease is stable and sufficiently controlled under treatment.
11. Any use of alcohol within 24 hours of admission to the clinic.
12. Plasma donation within 1 month of screening or any blood donation or corresponding blood loss during 3 months prior to screening.
13. Use of investigational agent within four weeks before Visit 1 or plans to initiate treatment with an investigational agent during the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female participants with suspected endometrial lesions
Enrollment: 8 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
MRI enhancing effect | Day 1
  MRI enhancing effect will be evaluated by assessing changes between pre-dose images and post-dose images acquired using longitudinal relaxation time (T1)-weighted imaging sequences, analysing contrast-to-noise in endometriosis lesions vs reference tissue, signal-to-noise in endometriosis lesions. Additional MR-scan characteristic parameters may be calculated if deemed appropriate.

SECONDARY OUTCOMES:
Diagnostic Value Evaluation for endometriosis lesions. | Day 1
  Compare the number, size and site of endometriosis lesions obtained by SN132D imaging to transvaginal ultrasound (TUS) and clinically used non-contrast MRI
Diagnostic Value Evaluation for deep pelvic endometriosis lesions. | Day 1
  Compare the number, size and site of deep pelvic endometriosis lesionsobtained by SN132D imaging to transvaginal ultrasound (TUS) and clinically used non-contrast MRI
Number of treatments related adverse events (AEs) | Day 1 up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ligita Jokubkiene, MD, PhD, Principal Investigator — Senior Consultant Skåne University Hospital, Assoc Prof Lund University
Locations (1):
- Kvinnokliniken, Skåne University Hospital, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No